CLINICAL TRIAL: NCT07109375
Title: Observational Prospective Cohort Study on Long-term Effective and Safe Use of Pegunigalsidase Alfa in Adult Fabry Patients Under "Real-world" Setting
Brief Title: Observational Study on Long-term Use of Pegunigalsidase Alfa in Fabry Patients in a Real-world Setting
Acronym: PEGASO
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi Italia (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: CHIT-2401
Record Dates: First submitted 2025-07-10; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Fabry Disease
Keywords: Pegunigalsidase alfa; Fabry disease; Real-world; Alpha-galactosidase A; Lysosomal storage disorders
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry patients: Adult patients whit genetically confirmed diagnosis of Fabry disease being treated or planning to start treatment with Pegunigalsidase alfa according to clinical practice. Participants will be required to meet the inclusion and exclusion criteria and sign informed consent to be enrolled in the study.
  Interventions: Drug: pegunigalsidase alfa

INTERVENTIONS:
Drug: pegunigalsidase alfa — Pegunigalsidase alfa is 2 mg/mL concentrate for solution and is administered via intravenous infusion every two weeks.
  Other Names: Elfabrio

SUMMARY:
PEGASO is an observational study designed to collect prospective data on the effectiveness and safety of pegunigalsidase alfa in adult patients with Fabry disease, being treated or planning to start treatment, under real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (≥ 18 years).
2. Patients with a clinical diagnosis of Fabry disease confirmed by α-Gal A assay and detection of mutation in α-Gal A gene.
3. Patients either taking or planning to take pegunigalsidase alfa as treatment for Fabry disease. The treatment decision must be made independently from participation in this study.
4. Written informed consent to participate in the study and for the processing of personal data.

Exclusion Criteria:

1. History of hypersensitivity reaction to pegunigalsidase alfa.
2. Presence of any medical, emotional, behavioural, or psychological condition that, in the judgment of the physician, could interfere with the ability to participate in the study.
3. Female subjects who are pregnant or planning to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients who have a genetically confirmed diagnosis of Fabry disease and are being treated or plan to initiate treatment with pegunigalsidase alfa as per clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of structural abnormalities of the left ventricle | 24 months
  Changes from baseline in structural abnormalities of the left ventricle assessed by echocardiography and defined by the presence of Left Ventricular Hypertrophy.
Assessment of left ventricular diastolic function | 12 and 24 months
  Changes from baseline in left ventricular diastolic function by echocardiography. Diastolic dysfunction will be assessed using early to late diastolic trans-mitral flow velocity.
Assessment of renal function | 6, 12, 18 and 24 months
  Changes from baseline in renal function by estimated Glomerular Filtration Rate.

SECONDARY OUTCOMES:
Assessment of peak oxygen uptake (pVO2) | 24 months
  Changes from baseline in peak oxygen uptake (pVO2) using cardiopulmonary exercise testing (CPET).
Assessment of carbon dioxide production (VCO2) | 24 months
  Changes from baseline in carbon dioxide production (VCO2) using cardiopulmonary exercise testing (CPET).
Assessment of NT-pro-BNP and high sensitivity cardiac troponin levels | 6, 12,18 and 24 months
  Changes from baseline in NT-pro-BNP and high sensitivity cardiac troponin levels.
Assessment of Cardiovascular Magnetic Resonance (CMR) | 12 and 24 months
  Changes from baseline in CMR assessed using T1 mapping to achieve myocardial tissue characterization.
Assessment of proteinuria and microalbuminuria | 6, 12, 18 and 24 months
  Changes from baseline in proteinuria and microalbuminuria assessed on 24-hour urine sample.
Assessment of Globotriaosylsphingosine (lyso-Gb3) | 3, 6, 12 and 24 months
  Changes from baseline in blood concentration of lyso-Gb3
Assessment of QoL outcomes using the Short Form Health Survey 36 (SF-36) | 12 and 24 months
  Changes from baseline in SF-36 score. It is a disease-specific questionnaire consisting of eight domains, each represented by a scale calculated as the weighted sum of responses in the respective sections. Each domain score ranges from 0 to 100, with all questions given equal weight. A score of 0 indicates the worst possible health status, while a score of 100 represents the best possible health status.
Assessment of QoL outcomes using the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 12 and 24 months
  Changes from baseline in KCCQ scores. It measures patient's perception of their health status, focusing on heart failure symptoms, the impact on physical and social functioning, and the overall effect of heart failure on their QoL within a 2-week recall period. It evaluates seven domains, with scores ranging from 0 to 100, where lower scores indicate more severe symptoms or limitations, while a score of 100 represents no symptoms, no limitations, and excellent quality of life.
Assessment of severity of neuropathic pain using Chronic Pain Grade (CPG) | 12 and 24 months
  Changes from baseline in CPG score. It is a 7-item questionnaire that evaluates chronic pain severity experienced over the past six months. Pain intensity is rated from 0 (no pain) to 10 ("pain as bad as it can be"). Scores for pain intensity and disability are combined to classify the overall severity of chronic pain into four grades, ranging from Grade 0 (no pain) to Grade IV (high disability, severely limiting).
Assessment of severity of neuropathic pain using Short Form of the Brief Pain Inventory (BPI-SF) | 12 and 24 months
  Changes from baseline in BPI-SF score. It is a 9-item questionnaire assessing Pain Intensity and Pain Interference, as its impact on daily functions, over the past 24 hours. Pain intensity is rated on a 0 (no pain) to 10 (pain as bad as you can imagine) scale, across four measures: worst, least, average, and current pain. Pain interference with daily activities is also scored from 0 (no interference) to 10 (completely interferes).
Assessment of gastrointestinal symptoms using the Gastrointestinal Symptoms Rating Scale (GSRS) | 12 and 24 months
  Changes from baseline in GSRS score. It is a 15-item questionnaire designed to assess changes in gastrointestinal symptoms across five clusters: reflux, abdominal pain, indigestion, diarrhea, and constipation. The GSRS uses a seven-point Likert-type scale, with scores ranging from 1 (no troublesome symptoms) to 7 (very troublesome symptoms).
Assessment of specific Fabry disease ocular findings | Baseline, 12 and 24 months
  Number of patients with presence of specific Fabry disease ocular findings (i.e. cornea verticillate) by slit lamp
Adverse events | 24 months
  Number of AEs
Adverse drug reactions to pegunigalsidase alfa | 24 months
  Number of ADRs
Anti-drug antibodies (ADAs) testing | 24 months
  Number of patients with ADAs
Infusion-Related Reactions (IRRs) | 24 months
  Number of patients and occurrence of IRRs

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pisani, MD, Principal Investigator — AOU Federico II, Dipartimento di Nefrologia, Napoli, Italy
Locations (1):
- AOU Federico II, Dipartimento di Nefrologia, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No